CLINICAL TRIAL: NCT00041275
Title: Randomized Double Blind Trial Of Megestrol Acetate Versus Placebo For The Treatment Of Inoperable Hepatocellular Carcinoma
Brief Title: Megestrol in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Medical Research Council (NMRC), Singapore (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000069460; NMRC-AHCC02; EU-20203
Record Dates: First submitted 2002-07-08; First posted 2003-01-28 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2002-09

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Megestrol Acetate

INTERVENTIONS:
Drug: megestrol acetate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of cancer cells. Hormone therapy using megestrol may fight liver cancer by blocking the uptake of estrogen. It is not yet known if megestrol is an effective treatment for liver cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of megestrol in treating patients who have liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with inoperable hepatocellular carcinoma treated with megestrol vs placebo.
* Compare the quality of life of patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral megestrol twice daily for 1 year.
* Arm II: Patients receive an oral placebo twice daily for 1 year. Quality of life is assessed at baseline and then monthly for 1 year.

PROJECTED ACCRUAL: A minimum of 300 patients (200 for arm I and 100 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC)

  * Histologically confirmed OR
  * Meets 2 of the following criteria:

    * Radiological evidence of HCC on CT scan, MRI, or ultrasound
    * Serum alpha-fetoprotein level at least 400 µg/L
    * Positive lipiodol retention
* Not amenable to surgery

PATIENT CHARACTERISTICS:

Age:

* 20 to 100

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 5.8 mg/dL

Renal:

* Creatinine less than 1.7 mg/dL

Other:

* Not pregnant
* No clinical encephalopathy
* No other malignancy within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemoembolization for HCC
* No prior systemic chemotherapy for HCC

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* No prior surgery for HCC

Other:

* No prior percutaneous injection for HCC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2002-05; Primary Completion 2007-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Survival measured weekly

SECONDARY OUTCOMES:
Quality of life as measured by EORTC quality of life instrument monthly

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, MBBS, FRCS, FAMS, Study Chair — National Cancer Centre, Singapore
Locations (12):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
- Yangon General Hospital, Yangon, Burma
- Rumah Sakit Sanglah, Denpasar, Bali, Indonesia
- Auckland City Hospital, Auckland, New Zealand
- Davao Doctors Hospital, Davao City, Philippines
- Singapore (2):
  - National Cancer Centre - Singapore, Singapore
  - Changi General Hospital, Singapore
- St. Vincent Hospital, Suwon, South Korea
- Chang-Gung Memorial Hospital - Taipei, Taipei, Taiwan
- Ramathibodi Hospital, Bangkok, Thailand
- Vietnam (2):
  - National Cancer Institute, Hà Nội
  - Cho Ray Hospital, Ho Chi Minh City

REFERENCES:
- [Result] Chow PK, Machin D, Chen Y, Zhang X, Win KM, Hoang HH, Nguyen BD, Jin MY, Lobo R, Findlay M, Lim CH, Tan SB, Gandhi M, Soo KC; Asia-Pacific Hepatocellular Carcinoma Trials Group. Randomised double-blind trial of megestrol acetate vs placebo in treatment-naive advanced hepatocellular carcinoma. Br J Cancer. 2011 Sep 27;105(7):945-52. doi: 10.1038/bjc.2011.333. Epub 2011 Aug 23. PMID 21863030